CLINICAL TRIAL: NCT00413270
Title: A Canadian Open-label, Multicenter, Expanded Access Study of Oral Nilotinib in Adult Patients With Imatinib-resistant or -Intolerant Chronic Myeloid Leukemia in Blast Crisis, Accelerated Phase, or Chronic Phase
Brief Title: Oral Nilotinib in Adults With Chronic Myeloid Leukemia (CML) in Blast Crisis Who Are Imatinib Resistant or Intolerant
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Other Study IDs: CAMN107ACA01
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Imatinib resistant,; Imatinib intolerant,; CML- blast crisis,; CML- Accelerated phase,; CML- chronic phase,; nilotinib,; Chronic myelogenous leukemia,; blast crisis,; accelerated phase,; chronic phase
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Blast Crisis | interventions — nilotinib

INTERVENTIONS:
Drug: nilotinib

SUMMARY:
This study will evaluate the safety of nilotinib in adult patients with imatinib-resistant or -intolerant CML-blast crisis, CML-accelerated phase or CML-chronic phase when treated with nilotinib. Patients will be provided access to nilotinib until the drug is available on the market.

ELIGIBILITY:
Inclusion Criteria:

* Imatinib resistant or intolerant Philadelphia chromosome positive CML in blast crisis
* Imatinib resistant or intolerant Philadelphia chromosome positive CML in accelerated phase
* Imatinib resistant or intolerant Philadelphia chromosome positive CML in chronic phase
* CML patients who have been treated with an investigational tyrosine kinase inhibitor who otherwise meet the definition of imatinib resistance or intolerance
* World Health Organization (WHO) performance status ≤ 2

Exclusion Criteria:

* Cytopathologically confirmed central nervous system (CNS) infiltration
* Impaired cardiac function
* Use of therapeutic coumarin derivatives
* Acute chronic liver or renal disease unrelated to tumor
* Other uncontrolled medical conditions
* Treatment with hematopoeitic colony stimulating factors
* Treatment with medications that have potential to prolong the QT interval
* Another malignancy currently clinically significant or requires active intervention

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- Canada (18):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Burnaby, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Oshawa, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Windsor, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan